CLINICAL TRIAL: NCT01099553
Title: Improving Bowel Preparation With an Education Video
Brief Title: Improving Bowel Preparation With an Educational Video
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Brian Jacobson, Associate Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-29152
Record Dates: First submitted 2010-04-02; First posted 2010-04-07 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Bowel Preparation
Keywords: Educational video; colonoscopy; bowel preparation; Bowel preparation for colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard preparation instructions (Other): The control arm will receive written instructions on preparing for a colonoscopy per standard of care at Boston Medical Center
  Interventions: Other: Written instructions
- Interventional (Experimental): The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus instructions asking them to watch an educational video on the Center for Digestive Disorders website
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Instructions to view an educational video about preparing for a colonoscopy
  Arms: Interventional
Other: Written instructions — Written instructions on preparing for a colonoscopy
  Arms: Standard preparation instructions

SUMMARY:
The investigators goal is to improve bowel preparations with an educational video on the Center for Digestive Disorders (CDD) website that explains the steps required for bowel preparation for those patients undergoing screening colonoscopies. The video will focus on explaining the purpose of a screening colonoscopy, the rationale for bowel preparation, the pre-colonoscopy diet, and the instructions for completing the laxative. In a randomized fashion, patients in the control group will receive the standard written bowel preparation instructions, while patients in the intervention group will receive standard written instructions plus a link to watch the instructional video. The investigators hypothesize that an educational tool that provides visual examples of a good and poor preparation, examples of the pre-colonoscopy diet, and an explanation of how to administer the laxative will lead to improved patient compliance and a better bowel preparation. In addition, the investigators hypothesize that a better quality bowel preparation will improve detection of colonic polyps and fewer recommendations for repeat colonoscopy based solely on inadequate bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* all outpatients
* age >18
* referred and scheduled for an elective screening colonoscopy

Exclusion Criteria:

* inpatients
* prisoners
* patients allergic to PEG-ELS based laxatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | Day of colonoscopy only
  The primary outcome will be the endoscopist's assessment of the quality of preparation using a standardized bowel preparation scale

SECONDARY OUTCOMES:
Histology of polyp | one week after colonoscopy
  number of adenomatous polyps
Colonoscope insertion and withdrawal times | Day of colonoscopy only
  time from insertion to cecum and time from cecum to anus
Patient compliance | Day of colonoscopy only
  Patient compliance with preparation instructions self-reported in a pre-procedure questionnaire
Preparation associated side effects | Day of colonoscopy only
  Presence and severity of preparation associated side effects including: blaoting, abdominal pain, and nausea/vomiting
Patient satisfaction | Day of colonoscopy only
  patient's perception of the helpfulness of the video as self-reported on a pre-procedure questionnaire.
Number of repeat colonoscopies due to inadequate bowel preparation | Day of colonoscopy only
  Blinded endoscopist's assesment about the need for a repeat colonoscopy due to inadequate bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Jacobson, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States